CLINICAL TRIAL: NCT07095829
Title: Development and Validation of a Prognostic Model of Postnatal Circulation in Fetuses With a Diagnosis of Pulmonary Atresia-critical Stenosis With Intact Ventricular Septum A Prospective Observational Cohort Study
Brief Title: Prognostic Model of Postnatal Circulation in Pulmonary Atresia-critical Stenosis With Intact Ventricular Septum
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Instituto de investigación Hospital 12 de Octubre (Unknown)
Responsible Party: Sponsor
Other Study IDs: PROGPAIVS
Record Dates: First submitted 2024-03-18; First posted 2025-07-31 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Atresia With Intact Ventricular Septum; Congenital Heart Disease; Fetal Cardiac Disorder
Keywords: Prognosis; Prenatal diagnosis; Ultrasound
MeSH Terms: conditions — Pulmonary Atresia with Intact Ventricular Septum; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective cohort: Retrospective cases that meet all the inclusion criteria and none of the exclusion criteria from 2013 until 2023 will be included for model development. They should be non-intervened cases in order to assess the natural history of the disease.
  Interventions: Other: No intervention
- Prospective cohort: Prospectively recruited cases will be included when meeting all the inclusion criteria and none of the exclusion ones. This cohort will serve as a validation cohort for the previously developed model. The nature of the study is observational. Clinicians will not be given the result of the model during the study and clinical practice will be routine.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Evaluation of natural history of the disease

SUMMARY:
Pulmonary atresia (PA)/critical stenosis (CS) with intact ventricular septum (PA/CS-IVS) is a rare congenital heart disease (CHD), that presents heterogeneously. Prognosis is conditioned by the possibility of achieving a primary repair with biventricular circulation (BV) or a one-and-a-half ventricle solution vs. a palliative approach bound to a univentricular (UV) circulation in which both survival and quality of life are significantly impaired. Predicting UV circulation prenatally is still a challenge.

The aim of this study is: 1/ to evaluate the natural history of the disease and develop a prognostic model for the prediction of transplantation-free survival with a biventricular or a one-and-a-half repair at 2 years postnatal age 2/ To develop a model to predict the risk of right ventricle dependent coronary circulation 3/ To evaluate prenatal and postnatal outcomes in non-intervened fetuses with a confirmed postnatal diagnosis of PA-CS/IVS including Intrauterine death, neonatal/Infant death, number of required postnatal procedures, need for oxygen support, need for cardiac transplantation

DETAILED DESCRIPTION:
This is an international retrospective and prospective observational cohort study including non-intervened fetuses with a diagnosis of PA-CS/IVS between 16+0 and 28+6 weeks of gestation.

A baseline fetal ultrasound examination will be recorded for all included cases. The primary aim of the study is to develop a prognostic and validate model for the type of postnatal circulation (transplantation-free survival with a biventricular or a one-and-a-half repair at 2 years postnatal age vs univentricular palliation or transplanted).

In order to maximize the number of included cases in this rare entity, the model will be developed on retrospective data from 2013 until 2023 and validated in a prospective cohort. Cases will be recruited in referral centers regardless of their offering of fetal pulmonary valvuloplasty. However, only non-prenatally-intervened cases will be used for analysis. Fetal and postnatal echocardiographic examinations will be reviewed by a core laboratory to confirm eligibility for inclusion and identify potential measurement errors.

Data from at least one fetal echo (the first diagnostic evaluation at the referral center) and one postnatal (the first one performed after birth) will be collected, each containing a comprehensive set of two-dimensional and Doppler measurements. Additionally, one additional follow-up scan performed at least 8 weeks apart from the baseline diagnostic scan (ideally between 28 and 32 weeks) will be included in the study as well. Analysis of the prenatal change of dimensions of the right heart structures and selected hemodynamic parameters will enable comparisons between centers regardless of off-protocol center-specific postnatal treatment policies.

ELIGIBILITY:
Inclusion Criteria:

* Absence of flow at the pulmonary valve (PA) or presence of thickened and domed. pulmonary valve cusps with a pinhole jet of flow.
* Doppler evidence of ductal-dependent pulmonary circulation.
* Intact ventricular septum.

Exclusion Criteria:

* Poor imaging windows and incomplete/poor quality scan
* Termination of pregnancy
* Cases initially included that undergo prenatal pulmonary valvuloplasty later on in pregnancy.
* Unconfirmed PA-CS/IVS at birth.
* Functional PA-CS/IVS (Ebstein malformation, monochorionic twins)
* Any associated cardiac defect except persistent left superior vena cava and aberrant right subclavian artery.
* Any significant (i.e that might influence outcome) extracardiac anomaly and/or known genetic syndromes. Also, if such a condition is present at inclusion but diagnosed only after birth, the case will be retrospectively excluded.

Ages: 16 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Screening data: All pregnant women with a fetus with suspected PA-CS/IVS will be screened for eligibility. If they meet all the inclusion criteria and none of the exclusion ones, they will be offered to participate. A complete count of screened, eligible, and included participants will be detailed in the final report of the study.
  Eligibility: As described in the next section, cases must meet all the inclusion criteria, and none of the exclusion ones.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Prediction of postnatal circulation | 3 years (1 recruitment, 2 follow-up)
  Transplantation-free survival with a non-univentricular circulation (biventricular or a one-and-a-half repair) at 2 years postnatal age: yes/no

SECONDARY OUTCOMES:
Prediction of coronary circulation | 3 years (1 recruitment, 2 follow-up)
  Prediction of right ventricle-dependent coronary circulation confirmed by cath or autopsy (yes/no)
Intrauterine death | 3 years (1 recruitment, 2 follow-up)
  Intrauterine death (yes/no)
Neonatal/Infant death in the first 2 years | 3 years (1 recruitment, 2 follow-up)
  Neonatal/Infant death in the first 2 years (yes/no)
Number of required postnatal surgical and catheter interventional procedure | 3 years (1 recruitment, 2 follow-up)
  Number of required postnatal surgical and catheter interventional procedures
Type of required postnatal surgical and catheter interventional procedures | 3 years (1 recruitment, 2 follow-up)
  Type of required postnatal surgical and catheter interventional procedures
O2 saturation at 30 days (%) | 3 years (1 recruitment, 2 follow-up)
  O2 saturation at 30 days (%)
Transplantation in the first two years | 3 years (1 recruitment, 2 follow-up)
  Transplantation in the first two years (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Villalaín González, MD PhD, Principal Investigator — Instituto de investigación imas12; Alberto Galindo Izquierdo, MD PhD, Principal Investigator — Instituto de investigación imas12
Locations (2):
- Hospital Universitario 12 de Octubre, Madrid, Spain
- University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT07095829/Prot_SAP_000.pdf